CLINICAL TRIAL: NCT03734081
Title: A First in Human (FIH) Study to Assess the Safety and Feasibility of the Bio-electrical One Day Capsule (ODC) System (Type 1 and 2 Capsules) in Overweight and Class 1 Obese Subjects
Brief Title: Safety and Feasibility Assessment of the Bio-electrical One Day Capsule System in Overweight and Class I Obese Participants
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The first cohort of 6 subjects that has been enrolled is being analyzed and evaluated on all safety parameters as described in the study protocol.
Sponsor: Melcap Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLD-012
Record Dates: First submitted 2018-11-04; First posted 2018-11-07 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2018-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gastric electrical stimulation with type 2 ODC (Experimental): Safety and feasibility assessment of the ODC system (type 2) capsule during and following gastric electrical stimulation protocol.
  Interventions: Device: ODC system (type 2 capsule)
- Electrical stimulation with type 2 ODC (Experimental): Safety and feasibility assessment of the ODC system (type 2) capsule during and following small and large bowel electrical stimulation protocol.
  Interventions: Device: ODC system (type 2 capsule)
- Electrical stimulation with type 1 ODC (Experimental): Safety and feasibility assessment of the ODC system (type 1 capsule) during and following small and large electrical stimulation protocol.
  Interventions: Device: ODC system (type 1 capsule)

INTERVENTIONS:
Device: ODC system (type 1 capsule) — ODC (one day capsule) type 1 is ingested by a subject and passes through the gastrointestinal tract. Electrical stimulation is the transferred from the capsule to the surrounding GI tissues. The capsule is excreted from the body through the intestinal tract in a natural manner with bowel movement.
  Arms: Electrical stimulation with type 1 ODC
Device: ODC system (type 2 capsule) — ODC (one day capsule) type 2 is ingested by a subject and passes through the gastrointestinal tract. Electrical stimulation is the transferred from the capsule to the surrounding GI tissues. The capsule is excreted from the body through the intestinal tract in a natural manner with bowel movement.
  Arms: Electrical stimulation with type 2 ODC; Gastric electrical stimulation with type 2 ODC

SUMMARY:
The study represents the first effort to prospectively investigate the Melcap's bio-electrical ingestible ODC system in human. The study goal is to evaluate the safety and feasibility of GES treatment in stomach and in the small and large bowel during and following the ingestion of the bio-electrical capsule under tight and controlled conditions.

DETAILED DESCRIPTION:
The problem of obesity in the adult population requires the exploration and development of new, safe and effective therapies to combat increasing growth. A novel Implantable Gastric Electrical Stimulation (GES), MEASTRO(R) Rechargeable System, has been recently approved by the American Food and Drug Administration (FDA) for use in weight reduction in patients aged 18 years through adulthood who have a Body Mass Index (BMI) of 40 to 45 kg/m2 with one or more obesity related co-morbid conditions, and have failed at least one supervised management program within the past 5 years.

Melcap System Ltd. has developed an innovative ingestible capsule system device that uses GES for the treatment of overweight and obesity. The system is intended to suppress hunger, reduce appetite, increase satiation and promote weight reduction in overweight and class I obese adults who have a Body Mass Index of 27 kg/m2 to 34.9 kg/m2 with no related co-morbid conditions.

The study is a FIH prospective, open label, randomized study. It will include a 3 days screening period and 4 days treatment session under a close supervision and follow up. Each subject will ingest a total of 2 capsules (ODC) on the first and the third day of the study. The total duration of subject participation including the termination visit will be eight days.

The study will be conducted at a single medical center, Meir Hospital, Israel.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 21-65 years old at time of screening
2. Body mass Index (BMI) >= 27 and <35
3. The subject has been under routine care of the investigator or another single physician that can supply a medical record for at least 4 months prior to enrollment
4. Female subjects at reproductive age that are tested negative for pregnancy
5. Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods during the whole study duration
6. No significant weight loss (<5%) within four months prior to enrollment (by self -report)
7. No recorded or treated psychological disorder(s) for at least six months prior to enrollment (by self report)
8. Not taking anti-depressant medication, for at least six months prior to enrollment.
9. Willingness to refrain from using prescription, over the counter or herbal weight loss products for the duration of he trial.
10. Personally motivated and willing to comply with all the requirements of the clinical trial
11. Able to understand, read and voluntary sign the inform consent form
12. Agree and able to sign the consent form for the Pillcam(R) patency capsule test as is in use at Meir MC.

Exclusion Criteria:

1. History o abdominal or gastrointestinal surgery (appendectomy, hernia repair, gynecological surgeries and cholecystectomy more than a year ago are allowed)
2. Prior bariatric surgery
3. Implanted electrical stimulation devices (e.g. pacemaker, defibrillator, neurostimulator)
4. Unwillingness to stop medication altering gastric pH and/or affecting GI motility during the entire study duration.
5. Known diagnosed psychiatric conditions that may impair subject's ability to comply with the study procedures (by self-report)
6. Use of anti-psychotic medications
7. Diagnosed with an eating disorder including bulimia and binge eating
8. Swallowing difficulties
9. Significant active or unstable acute or chronic illnesses/ diseases including gastrointestinal, systemic (non-gastrointestinal) and psychiatric conditions
10. Use of another investigation device or agent in the 30 days prior to enrollment
11. Women who are pregnant, lactating or anticipate to becoming pregnant within the study duration
12. Planned or contemplated use of Magnetic Resonance Imaging (MRI) or any (e.g. oncologic) radiation during the course of the trial.
13. Have a family member who is currently participating in this clinical trial
14. Any other conditions that, in the opinion of the investigator, would make the subject unsuitable for the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of all adverse events | During the whole study duration (approximately 8 days)
  Safety evaluation
Incidence of device-related adverse events | During the whole study duration (approximately 8 days)
  Safety evaluation
Incidence of clinically significant abnormal laboratory values as determined by the investigator | During the whole study duration (approximately 8 days)
  Safety evaluation
Excretion of the study capsules in a natural manner | up to 3 days after the days of the capsules ingestion
  Safety evaluation - confirmation of the capsule excretion from the body

SECONDARY OUTCOMES:
Satiety levels | Day #1 and #3 of the treatment period
  Changes in satiety levels resulting of the electrical stimulation
Appetite levels | Day #1 and #3 of the treatment period
  Changes in appetite levels resulting of the electrical stimulation
Postprandial symptoms | Day #1, #2, #3 and #4 of the treatment period
  Evaluation of postprandial symptoms during the treatment period
Response to nutrient drink test | Day #3 of the screening period and and day #4 of the treatment period
  Determination of the maximum tolerable drinking volume followed by postprandial symptoms measurement
Appetite-related hormone | Day #1 and Day #3 of the treatment period
  Evaluation of appetite- related hormones levels change as a result of the stimulation applied

CONTACTS AND LOCATIONS:
Overall Officials: Timna Naftali, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No